CLINICAL TRIAL: NCT03848832
Title: A Randomized, Double-blind, Placebo-controlled Trial to Investigate the Efficacy and Safety of Cannabidiol Oral Solution (GWP42003-P, CBD-OS) in Patients With Rett Syndrome
Brief Title: Efficacy and Safety of Cannabidiol Oral Solution (GWP42003-P, CBD-OS) in Patients With Rett Syndrome
Acronym: ARCH
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The study was terminated due to enrollment challenges and the COVID-19 pandemic.
Sponsor: Jazz Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GWND18064; 2018-003370-27 (EudraCT Number)
Record Dates: First submitted 2019-02-19; First posted 2019-02-21 (Actual); Results first posted 2021-12-29 (Actual); Last update posted 2022-09-02 (Actual); Status verified 2022-08

CONDITIONS: Rett Syndrome; RTT
Keywords: Cannabidiol; CBD; Epidiolex; GWP42003-P
MeSH Terms: conditions — Rett Syndrome | interventions — Cannabidiol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- 5 milligrams per kilogram per day (mg/kg/day) GWP42003-P (Experimental): 100 milligrams per milliliter (mg/mL) GWP42003-P oral solution. Taken twice daily (morning and evening).
  Interventions: Drug: GWP42003-P
- 15 mg/kg/day GWP42003-P (Experimental): 100 mg/mL GWP42003-P oral solution. Taken twice daily (morning and evening).
  Interventions: Drug: GWP42003-P
- Placebo (Placebo Comparator): Placebo oral solution (0 mg/mL GWP42003-P) volume matched to 5 mg/kg/day or 15 mg/kg/day GWP42003-P. Taken twice daily (morning and evening).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GWP42003-P — GWP42003-P presented as an oral solution containing cannabidiol
  Other Names: Cannabidiol; CBD; Epidiolex; CBD-OS
  Arms: 15 mg/kg/day GWP42003-P; 5 milligrams per kilogram per day (mg/kg/day) GWP42003-P
Drug: Placebo — Matching placebo oral solution
  Arms: Placebo

SUMMARY:
To evaluate the efficacy of cannabidiol oral solution (GWP42003-P, CBD-OS) in reducing symptom severity when compared with placebo, in participants with Rett syndrome.

ELIGIBILITY:
Key Inclusion Criteria:

* Participant (if possessing adequate understanding, in the investigator's opinion) and/or their parent(s)/legal representative is willing and able to give informed consent/assent for participation in the trial.
* Participant and their caregiver are willing and able (in the investigator's opinion) to comply with all trial requirements (including the completion of all caregiver assessments by the same caregiver throughout the trial).
* Participant must weigh at least 10 kilograms.
* Clinical diagnosis of Rett syndrome (typical or atypical), defined according to RettSearch Consortium criteria
* Confirmed pathogenic genetic mutation of the MECP2 gene
* Participant must be post-regression (≥ 6 months since last loss of hand use or verbal language or gross motor regression).
* Participant must have a disease severity of between 10 and 36, defined according to the Clinical Severity Scale (CSS).
* All medications or interventions (including antiepileptic drugs [AEDs] and non-pharmacological interventions - dietary supplements, probiotics, physical therapy, speech therapy, etc.) for Rett syndrome-related symptoms must have been stable for 4 weeks prior to screening and the participant/caregiver must be willing to maintain a stable regimen throughout the trial.
* Ability to swallow the investigational medicinal product (IMP) provided as a liquid solution, or the ability for IMP to be delivered via gastrostomy (G) or nasogastric (NG) feeding tube (only G-or NG-tubes made from polyurethane or silicon are allowed)
* Participant and/or parent(s)/legal representative is willing to allow the responsible authorities to be notified of participation in the trial, if mandated by local law.
* Participant and/or parent(s)/legal representative is willing to allow the participant's primary care practitioner (if they have one) and consultant (if they have one) to be notified of participation in the trial, if the primary care practitioner/consultant is different than the investigator.

Key Exclusion Criteria:

* Participant meets exclusion criteria for Rett syndrome diagnosis (traumatic brain injury, neurometabolic disease, or severe infection that causes neurological problems; grossly abnormal psychomotor development in the first 6 months of life).
* Participant has clinically significant abnormal laboratory values, in the investigator's opinion.
* Participant is taking more than 2 concurrent AEDs.
* Any history of suicidal behavior or any suicidal ideation in the last month or at screening
* Clinically relevant abnormalities in the electrocardiogram (ECG) measured at screening or randomization
* Concurrent cardiovascular conditions which will, in the investigator's opinion, interfere with the ability to assess their ECGs or put the participant at risk because of participation in the trial
* First or second degree relative with a history of significant ECG abnormalities, in the opinion of the investigator (e.g. premature cardiac arrest, sudden death)
* Any known or suspected hypersensitivity to cannabinoids or any of the excipients of the IMP (active or placebo), such as sesame oil
* Participant has moderately impaired hepatic function at screening, defined as alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > 3 × upper limit of normal (ULN) or total bilirubin > 2 × ULN.
* Participant is of childbearing potential, unless willing to ensure that they or their partner use a highly effective method of birth control (e.g., combined [estrogen and progestogen containing] hormonal contraception associated with inhibition of ovulation [oral, intravaginal, or transdermal], progestogen-only hormonal contraception associated with inhibition of ovulation [oral, injectable, or implantable], intrauterine devices/hormone-releasing systems, bilateral tubal occlusion, vasectomized partner, sexual abstinence) during the trial and for 3 months thereafter.
* Pregnant (positive pregnancy test) or lactating
* Received an IMP within the 3 months prior to screening
* Participant has been taking felbamate for less than 1 year prior to screening.
* Currently using or has used recreational or medicinal cannabis, cannabinoid-based medications (including Sativex®), or cannabidiol oral solutions (including CBD-OS [GWP42003-P]) within the 3 months prior to screening and is unwilling to abstain for the duration of the trial
* Participant has a positive delta-9-tetrahydrocannabinol (THC) test at screening.
* Any other systemic dysfunction (e.g., gastrointestinal, renal, respiratory) or significant disease or disorder which, in the opinion of the investigator, may either put the participant at risk because of participation in the trial, may influence the result of the trial, or the participant's ability to participate in the trial
* Any abnormalities identified following a physical examination of the participant that, in the opinion of the investigator, would jeopardize the safety of the participant if she took part in the trial
* Participant has been previously randomized into this trial.
* Participant has traveled outside the country of residence planned during the trial.

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 29 (Actual)
Dates: Start 2019-07-29 (Actual); Primary Completion 2021-01-21 (Actual); Study Completion 2021-01-21 (Actual)

CONTACTS AND LOCATIONS:
Locations (23):
- United States (14):
  - Clinical Trial Site, Birmingham, Alabama
  - Clinical Trial Site, San Diego, California
  - Clinical Trial Site, Aurora, Colorado
  - Clinical Trial Site, Chicago, Illinois
  - Clinical Trial Site, Baltimore, Maryland
  - Clinical Trial Site, Boston, Massachusetts
  - Clinical Trial Site, Saint Paul, Minnesota
  - Clinical Trial Site, St Louis, Missouri
  - Clinical Trial Site, The Bronx, New York
  - Clinical Trial Site, Cincinnati, Ohio
  - Clinical Trial Site, Philadelphia, Pennsylvania
  - Clinical Trial Site, Greenwood, South Carolina
  - Clinical Trial Site, Nashville, Tennessee
  - Clinical Trial Site, Houston, Texas
- Italy (4):
  - Clinical Trial Site, Genoa
  - Clinical Trial Site, Messina
  - Clinical Trial Site, Milan
  - Clinical Trial Site, Rome
- Spain (3):
  - Clinical Trial Site, Barcelona
  - Clinical Trial Site, Madrid
  - Clinical Trial Site, Valencia
- United Kingdom (2):
  - Clinical Trial Site, Liverpool
  - Clinical Trial Site, London

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 41 participants were screened for eligibility; 29 were randomized to the study treatments, and 12 were screen failures.
Groups:
- 5 mg/kg/Day GWP42003-P: Participants received 5 milligrams (mg)/kilogram (kg)/day GWP42003-P, administered as 100 mg/milliliter (mL) oral solution twice daily (BID).
- 15 mg/kg/Day GWP42003-P: Participants received 15 mg/kg/day GWP42003-P, administered as 100 mg/mL oral solution BID.
- Placebo: Participants received placebo oral solution matched to 5 or 15 mg/kg/day GWP42003-P, BID.
Period: Overall Study
Arm/Group | 5 mg/kg/Day GWP42003-P | 15 mg/kg/Day GWP42003-P | Placebo
Started | 10 | 9 | 10
Completed | 7 | 6 | 4
Not Completed | 3 | 3 | 6
Not completed — Withdrawal of Consent Due To Covid-19 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 1
Not completed — Withdrawal (Covid-19) | 0 | 2 | 0
Not completed — Physician Decision | 2 | 1 | 3
Not completed — Sponsor Decision - Covid-19 Precaution | 0 | 0 | 1
Not completed — Adverse Event | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: One participant assigned to the 5 mg/kg/Day placebo group was misdosed with 5 mg/kg/Day GWP42003-P. The participant was included in the 5 mg/kg/Day placebo group in the Intent-to-Treat Set but was included in the 5 mg/kg/day GWP42003-P group in the Safety Analysis Set (for which Baseline data are reported).
Groups:
- Total: Total of all reporting groups
Arm/Group | 5 mg/kg/Day GWP42003-P | 15 mg/kg/Day GWP42003-P | Placebo | Total
Number analyzed (Participants) | 11 | 9 | 9 | 29
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 11 | 9 | 9 | 29
  Between 18 and 65 years | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 9.7 (6.02) | 10.7 (3.64) | 8.6 (5.53) | 9.7 (5.11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 9 | 9 | 29
  Male | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 1
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 10 | 9 | 9 | 28
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Mean Rett Syndrome Behaviour Questionnaire (RSBQ) Total Score at Week 24 for the 15 mg/kg/Day GWP42003-P Dose Level Compared With Placebo
Description: RSBQ is a caregiver-completed questionnaire that measures the frequency of current disease characteristics (45 items) in individuals with Rett Syndrome. Each item is rated on a 3-point scale (0-2); 0 indicating an item that is "not true as far as you know," 1 indicating an item is "somewhat or sometimes true," and 2 indicating an item that is "very true or often true." Item 31 ("Uses eye gaze to convey feelings, needs and wishes") is reverse scored (0 indicating "very true or often true", 1 indicating "somewhat or sometimes true," and 2 indicating "not true as far as you know"). The total summed score ranges from 0 to 90, with higher scores representing greater severity.
Time Frame: Baseline; Week 24
Population: Intent-to-Treat (ITT) Set: All randomized participants who received at least 1 dose of drug in the trial, and had Baseline efficacy data. Participants with non-missing data were included for analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 15 mg/kg/Day GWP42003-P | Placebo
Number analyzed (Participants) | 9 | 10
units on a scale
  Baseline | 45.9 (16.77) | 50.0 (7.56)
  Change from Baseline at Week 24: number analyzed (Participants) | 7 | 7
  Change from Baseline at Week 24 | -12.1 (13.63) | -6.1 (7.22)

2. Secondary Outcome: Change From Baseline in the Mean RSBQ Total Score at Week 24 for the 5 mg/kg/Day GWP42003-P Dose Level Compared With Placebo
Description: RSBQ is a caregiver-completed questionnaire that measures the frequency of current disease characteristics (45 items) in individuals with Rett Syndrome. Each item is rated on a 3-point scale (0-2); 0 indicating an item that is "not true as far as you know," 1 indicating an item is "somewhat or sometimes true," and 2 indicating an item that is "very true or often true." Item 31 ("Uses eye gaze to convey feelings, needs and wishes") is reverse scored (0 indicating "very true or often true", 1 indicating "somewhat or sometimes true," and 2 indicating "not true as far as you know"). The total summed score ranges from 0 to 90, with higher scores represent greater severity.
Time Frame: Baseline; Week 24
Population: ITT Set. Participants with non-missing data were included for analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 5 mg/kg/Day GWP42003-P | Placebo
Number analyzed (Participants) | 10 | 10
units on a scale
  Baseline | 39.8 (12.80) | 50.0 (7.56)
  Change from Baseline at Week 24: number analyzed (Participants) | 9 | 7
  Change from Baseline at Week 24 | 0.4 (12.51) | -6.1 (7.22)

3. Secondary Outcome: Mean Clinical Global Impressions - Improvement (CGI-I) Score at Week 24
Description: CGI-I is a 7-point scale that requires the clinician to assess how much a participant's illness has improved or worsened relative to a Baseline state at the beginning of the intervention. This is rated as: 1 = very much improved; 2 = much improved; 3 = minimally improved; 4 = no change; 5 = minimally worse; 6 = much worse; or 7 = very much worse.
Time Frame: Baseline; Week 24
Population: ITT Set. Participants with non-missing data were included for analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 5 mg/kg/Day GWP42003-P | 15 mg/kg/Day GWP42003-P | Placebo
Number analyzed (Participants) | 10 | 9 | 10
units on a scale | 3.2 (1.20) | 2.9 (1.07) | 3.1 (0.38)

4. Secondary Outcome: Change From Baseline in Mean Clinician Global Impressions - Severity (CGI-S) Score at Week 24
Description: CGI-S is a 7-point scale that requires the clinician to rate the severity of the participant's illness at the time of assessment relative to the clinician's experience with participants who had the same diagnosis. This is rated as: 1 = normal, not at all ill; 2 = borderline ill; 3 = mildly ill; 4 = moderately ill; 5 = markedly ill; 6 = severely ill; or 7 = extremely ill.
Time Frame: Baseline; Week 24
Population: ITT Set. Participants with non-missing data were included for analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 5 mg/kg/Day GWP42003-P | 15 mg/kg/Day GWP42003-P | Placebo
Number analyzed (Participants) | 10 | 9 | 10
units on a scale
  Baseline | 4.3 (1.25) | 4.2 (0.67) | 4.4 (0.84)
  Change from Baseline at Week 24: number analyzed (Participants) | 9 | 7 | 7
  Change from Baseline at Week 24 | -0.1 (0.33) | -0.1 (0.38) | 0.0 (0.00)

5. Secondary Outcome: Change From Baseline in Mean RSBQ Subscale Scores at Week 24
Description: RSBQ is a caregiver-completed questionnaire that measures the frequency of current disease characteristics in individuals with Rett Syndrome. The 45-item RSBQ is comprised of 8 subscales: 1) general mood (score range 0-16), 2) breathing problems (range 0-10), 3) hand behaviors (range 0-12), 4) face movements (range 0-8), 5) body rocking (BR)/expressionless face (range 0-12), 6) night-time behaviors (range 0-6), 7) anxiety/fear (range 0-8), 8) walking/standing (range 0-4). Each item is rated on a 3-point scale (0-2); 0 indicating an item that is "not true as far as you know," 1 indicating an item is "somewhat or sometimes true," and 2 indicating an item that is "very true or often true." Item 31 ("Uses eye gaze to convey feelings, needs and wishes") is reverse scored (0 indicating "very true or often true", 1 indicating "somewhat or sometimes true," and 2 indicating "not true as far as you know"). Higher scores representing greater severity. CFB = Change from Baseline.
Time Frame: Baseline; Week 24
Population: ITT Set. Participants with non-missing data were included for analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 5 mg/kg/Day GWP42003-P | 15 mg/kg/Day GWP42003-P | Placebo
Number analyzed (Participants) | 10 | 9 | 10
units on a scale
  Baseline General Mood Score | 6.0 (3.65) | 8.2 (4.58) | 8.9 (3.14)
  CFB General Mood Score: number analyzed (Participants) | 9 | 7 | 7
  CFB General Mood Score | -0.6 (2.70) | -4.9 (2.67) | -2.6 (2.57)
  Baseline Breathing Problems Score | 4.7 (2.45) | 5.0 (3.08) | 5.0 (3.43)
  CFB Breathing Problems Score: number analyzed (Participants) | 9 | 7 | 7
  CFB Breathing Problems Score | 0.2 (1.86) | -1.0 (1.53) | -0.3 (1.25)
  Baseline Hand Behaviors Score | 7.8 (2.15) | 7.6 (3.54) | 9.1 (2.08)
  CFB Hand Behaviors Score: number analyzed (Participants) | 9 | 7 | 7
  CFB Hand Behaviors Score | 0.7 (2.24) | -0.9 (3.29) | 0.1 (0.90)
  Baseline Face Movements Score | 2.3 (2.45) | 4.6 (2.13) | 4.3 (2.21)
  CFB Face Movements Score: number analyzed (Participants) | 9 | 7 | 7
  CFB Face Movements Score | 0.0 (1.12) | -1.4 (1.72) | -0.1 (1.07)
  Baseline Body Rocking/Expressionless Face Score | 4.5 (2.59) | 5.1 (1.96) | 5.4 (2.59)
  CFB Body Rocking/Expressionless Face Score: number analyzed (Participants) | 9 | 7 | 7
  CFB Body Rocking/Expressionless Face Score | 0.6 (2.46) | -0.6 (1.13) | -0.1 (1.86)
  Baseline Night-time Behaviors Score | 0.8 (1.14) | 0.8 (0.97) | 1.8 (1.69)
  CFB Night-time Behaviors Score: number analyzed (Participants) | 9 | 7 | 7
  CFB Night-time Behaviors Score | 0.2 (0.97) | -0.1 (1.46) | -0.3 (1.11)
  Baseline Anxiety/Fear Score | 4.0 (1.89) | 4.6 (2.46) | 5.1 (1.45)
  CFB Anxiety/Fear Score: number analyzed (Participants) | 9 | 7 | 7
  CFB Anxiety/Fear Score | -0.2 (1.92) | -1.3 (2.29) | -1.7 (0.95)
  Baseline Walking/Standing Score | 2.7 (1.64) | 2.1 (1.36) | 2.9 (1.29)
  CFB Walking/Standing Score: number analyzed (Participants) | 9 | 7 | 7
  CFB Walking/Standing Score | 0.9 (2.09) | 0.0 (0.58) | 0.1 (1.07)

6. Secondary Outcome: Change From Baseline in Mean 9-items Motor Behavioral Assessment (MBA-9) Total Score and Subscale Scores at Week 24
Description: MBA-9 is derived from the full MBA scale (37 Rett syndrome symptoms) by selecting the items deemed amenable to change and which reflected areas of meaningful clinical change. the MBA-9 includes 9 items (1-Regression of motor skills; 2-Poor eye/social contact; 3-Lack of sustained interest; 4-Does not reach for objects or people; 5-Chewing difficulties; 6-Speech disturbance; 7-Hand clumsiness; 8-Dystonia and 9-Hypertonia/rigidity); for each item, the severity of current symptoms is rated by the investigator on a 5-point numerical scale ranging from 0 to 4 with higher scores representing greater severity (0 = normal or never; 1 = mild or rare; 2 = moderate or occasional; 3 = marked or frequent; 4 = very severe or constant). Total MBA-9 score was calculated by summing the scores of 9 different subscale items. The total summed score ranges from 0 to 36, with higher scores representing greater severity. CFB = Change from Baseline.
Time Frame: Baseline; Week 24
Population: ITT Set. Participants with non-missing data were included for analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 5 mg/kg/Day GWP42003-P | 15 mg/kg/Day GWP42003-P | Placebo
Number analyzed (Participants) | 10 | 9 | 10
units on a scale
  Baseline Regression of Motor Skills | 2.2 (1.23) | 2.6 (0.88) | 2.6 (0.84)
  CFB Regression of Motor Skills: number analyzed (Participants) | 9 | 7 | 7
  CFB Regression of Motor Skills | 0.3 (1.58) | -0.3 (0.49) | 0.0 (0.58)
  Baseline Poor Eye/Social Contact | 1.7 (0.82) | 1.6 (1.01) | 1.5 (0.97)
  CFB Poor Eye/Social Contact: number analyzed (Participants) | 9 | 7 | 7
  CFB Poor Eye/Social Contact | 0.0 (0.87) | -0.1 (0.69) | -0.9 (1.07)
  Baseline Lack of Sustained Interest | 1.8 (0.79) | 2.1 (1.17) | 1.5 (0.71)
  CFB Lack of Sustained Interest: number analyzed (Participants) | 9 | 7 | 7
  CFB Lack of Sustained Interest | 0.0 (0.71) | -0.3 (1.11) | -0.1 (0.38)
  Baseline Does Not Reach for Objects or People | 2.0 (1.25) | 1.9 (1.05) | 2.3 (1.25)
  CFB Does Not Reach for Objects or People: number analyzed (Participants) | 9 | 7 | 7
  CFB Does Not Reach for Objects or People | -0.4 (2.24) | -0.4 (0.98) | 0.1 (1.21)
  Baseline Chewing Difficulties | 1.3 (1.34) | 1.3 (0.50) | 1.1 (0.74)
  CFB Chewing Difficulties: number analyzed (Participants) | 9 | 7 | 7
  CFB Chewing Difficulties | -0.2 (0.67) | 0.0 (0.00) | 0.4 (0.53)
  Baseline Speech Disturbance | 3.0 (0.47) | 2.8 (0.83) | 2.7 (0.48)
  CFB Speech Disturbance: number analyzed (Participants) | 9 | 7 | 7
  CFB Speech Disturbance | 0.0 (0.00) | 0.0 (0.58) | 0.3 (0.49)
  Baseline Hand Clumsiness | 2.8 (1.14) | 2.8 (1.56) | 3.1 (1.10)
  CFB Hand Clumsiness: number analyzed (Participants) | 9 | 7 | 7
  CFB Hand Clumsiness | -0.6 (1.33) | -0.4 (1.13) | 0.0 (0.58)
  Baseline Dysonia | 1.0 (1.41) | 1.2 (1.56) | 1.0 (1.41)
  CFB Dysonia: number analyzed (Participants) | 9 | 7 | 7
  CFB Dysonia | 0.4 (1.42) | -0.1 (0.90) | 0.1 (1.46)
  Baseline Hypertonia/Rigidity | 1.4 (1.51) | 1.1 (1.45) | 1.0 (1.41)
  CFB Hypertonia/Rigidity: number analyzed (Participants) | 9 | 7 | 7
  CFB Hypertonia/Rigidity | 0.4 (0.73) | -0.1 (0.38) | 0.0 (1.00)
  Baseline MBA-9 Total Score | 17.2 (5.81) | 17.3 (6.78) | 16.8 (5.96)
  CFB MBA-9 Total Score: number analyzed (Participants) | 9 | 7 | 7
  CFB MBA-9 Total Score | 0.0 (4.87) | -1.9 (4.06) | 0.0 (3.92)

7. Secondary Outcome: Change From Baseline in Mean Children's Sleep Habits Questionnaire (CSHQ) Total Score and Subscale Scores at Week 24
Description: CSHQ is a caregiver-completed sleep screening instrument designed for school-aged children; which includes 33 items within 8 subscales: 1) bedtime resistance (score range 6-18), 2) sleep onset delay (range 1-3), 3) sleep duration (range 3-9), 4) sleep anxiety (range 4-12), 5) night wakings (range 3-9), 6) parasomnias (range 7-21), 7) sleep-disordered breathing (range 3-9), 8) daytime sleepiness (range 8-24). Item scores range from 1 to 3, where 3="usually" (≥5 times/week), 2="sometimes" (2-4 times/week), and 1="rarely" (≤1 time/week); for items 31 and 32; 3=fall asleep, 2=very sleepy, 1=not sleepy. In general, a score of 3 indicates greater severity, however, 6 items (1-Goes to bed at same time; 2-Falls asleep in 20 minutes; 3-Falls asleep in own bed; 10-Sleeps the right amount; 11-Sleeps same amount each day; 26-Wakes by himself) are reverse scored. Total summed score ranges from 33 to 99, with higher scores representing more disturbed sleep behavior. CFB = Change from Baseline.
Time Frame: Baseline; Week 24
Population: ITT Set. Participants with non-missing data were included for analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 5 mg/kg/Day GWP42003-P | 15 mg/kg/Day GWP42003-P | Placebo
Number analyzed (Participants) | 10 | 9 | 10
units on a scale
  Baseline Total Score | 49.8 (9.75) | 46.7 (4.90) | 49.4 (5.42)
  CFB Total score: number analyzed (Participants) | 9 | 7 | 7
  CFB Total score | -1.6 (6.17) | -5.0 (6.14) | -3.7 (4.07)
  Baseline Bedtime resistance | 9.2 (3.43) | 7.3 (2.12) | 7.0 (1.25)
  CFB Bedtime resistance: number analyzed (Participants) | 9 | 7 | 7
  CFB Bedtime resistance | 0.0 (1.00) | -0.4 (1.27) | -0.1 (1.68)
  Baseline Sleep onset delay | 1.5 (0.71) | 1.4 (0.53) | 1.8 (0.79)
  CFB Sleep onset delay: number analyzed (Participants) | 9 | 7 | 7
  CFB Sleep onset delay | 0.1 (1.27) | -0.1 (0.69) | -0.6 (0.53)
  Baseline Sleep duration | 4.7 (2.41) | 3.4 (0.73) | 4.5 (1.58)
  CFB Sleep duration: number analyzed (Participants) | 9 | 7 | 7
  CFB Sleep duration | 0.4 (1.13) | -0.3 (0.95) | -0.4 (1.72)
  Baseline Sleep anxiety | 5.6 (1.65) | 4.6 (0.73) | 4.9 (1.10)
  CFB Sleep anxiety: number analyzed (Participants) | 9 | 7 | 7
  CFB Sleep anxiety | -0.1 (0.78) | -0.1 (0.38) | 0.0 (1.15)
  Baseline Night wakings | 5.3 (2.36) | 4.4 (1.33) | 4.6 (1.43)
  CFB Night wakings: number analyzed (Participants) | 9 | 7 | 7
  CFB Night wakings | -0.4 (0.88) | -0.6 (1.40) | 0.1 (0.69)
  Baseline Parasomnias | 11.0 (1.49) | 10.4 (1.42) | 11.7 (2.63)
  CFB Parasomnias: number analyzed (Participants) | 9 | 7 | 7
  CFB Parasomnias | -0.6 (1.51) | -1.1 (1.68) | -1.4 (2.30)
  Baseline Sleep disordered breathing | 4.2 (1.69) | 4.0 (1.22) | 3.7 (1.06)
  CFB Sleep disordered breathing: number analyzed (Participants) | 9 | 7 | 7
  CFB Sleep disordered breathing | -0.4 (1.74) | -0.9 (1.07) | -0.1 (0.38)
  Baseline Daytime sleepiness | 11.6 (3.20) | 13.2 (2.39) | 13.7 (2.50)
  CFB Daytime sleepiness: number analyzed (Participants) | 9 | 7 | 7
  CFB Daytime sleepiness | -0.7 (3.64) | -1.4 (2.07) | -1.3 (2.56)

ADVERSE EVENTS:
Time Frame: Up to approximately 207 days
Description: Safety Analysis Set: All participants who received at least 1 dose of investigational medicinal product in the trial were included and analyzed according to the treatment received. One participant who was assigned to the placebo group received GWP42003-P 5 mg/kg. For safety analyses, this participant was assigned to the GWP42003-P 5 mg/kg group.
Arm/Group | 5 mg/kg/Day GWP42003-P | 15 mg/kg/Day GWP42003-P | Placebo
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/9 | 0/9
Serious Adverse Events (participants affected / at risk) | 2/11 | 2/9 | 1/9
Other Adverse Events (participants affected / at risk) | 9/11 | 7/9 | 7/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 5 mg/kg/Day GWP42003-P (N=11) | 15 mg/kg/Day GWP42003-P (N=9) | Placebo (N=9)
COVID-19 (Infections and infestations) | 1 (1) | 1 (1) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Dyskinesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 5 mg/kg/Day GWP42003-P (N=11) | 15 mg/kg/Day GWP42003-P (N=9) | Placebo (N=9)
Coagulopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Eosinophilia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Macrocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1)
Ocular hyperaemia (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 2 (2) | 0 (0)
Faeces soft (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Tooth discolouration (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 2 (3) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 2 (3) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 2 (2) | 0 (0) | 1 (2)
Otitis media (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pharyngitis streptococcal (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 3 (5)
Viral upper respiratory tract infection (Infections and infestations) | 1 (4) | 0 (0) | 0 (0)
Sunburn (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Blood thyroid stimulating hormone increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Breath sounds abnormal (Investigations) | 0 (0) | 1 (1) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Mean cell volume increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Selenium deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Joint stiffness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Scoliosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Balance disorder (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Disturbance in attention (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0)
Dizziness postural (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Drooling (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Hyperreflexia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Lethargy (Nervous system disorders) | 0 (0) | 3 (3) | 0 (0)
Seizure (Nervous system disorders) | 1 (2) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Agitation (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Bruxism (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Dermatillomania (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 2 (2)
Irritability (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Middle insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Nervousness (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Sleep disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Choking (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 1 (1)
Skin discolouration (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
This study was terminated early due to enrollment challenges and the Coronavirus disease-2019 (COVID-19) pandemic. Numbers of participants in each treatment groups were small, which precluded the planned formal statistical inferences and limited data interpretation.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2020-08-07): https://cdn.clinicaltrials.gov/large-docs/32/NCT03848832/Prot_000.pdf
  • Statistical Analysis Plan (2021-03-31): https://cdn.clinicaltrials.gov/large-docs/32/NCT03848832/SAP_001.pdf